CLINICAL TRIAL: NCT03387904
Title: A Randomized, Eploratory, Open Clinical Trial to Compare the Efficacy and Safety of Anlotinib Plus Irinotecan Versus Irinotecan in Patients With Esophageal Squamous Cell Carcinoma
Brief Title: Study of Anlotinib Plus Irinotecan in Patients With Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-11-II-01
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Anlotinib
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — anlotinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anlotinib Plus Irinotecan (Experimental): Anlotinib QD po.and Irinotecan Day 1,8 ivgtt. Both should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib Plus Irinotecan
- Irinotecan (Active Comparator): Irinotecan Day 1,8 ivgtt and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Anlotinib Plus Irinotecan — Anlotinib QD po.and Irinotecan Day 1,8 ivgtt.
  Arms: Anlotinib Plus Irinotecan
Drug: Irinotecan — Irinotecan Day 1,8 ivgtt
  Arms: Irinotecan

SUMMARY:
To compare the effects and safety of Anlotinib Plus Irinotecan versus Irinotecan in patients with esophageal squamous cell carcinoma(ESCC).

DETAILED DESCRIPTION:
In recent years, anti-angiogenic therapy has made some progress in the treatment of advanced esophageal squamous cell carcinoma.In clinical use, the efficacy of antiangiogenic monotherapy was low, with a median progression-free survival (PFS) of only 3 to 4 months.We conducted a randomized, open clinical Trial to evaluate efficacy and safety of anlotinib hydrochloride combined with irinotecan versus irinotecan monotherapy in patients with advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of esophageal squamous cell carcinoma;
* At least one measurable lesion (by RECIST1.1);
* Patients who have failed to a chemoradiation treatment;
* 18-75，ECOG PS:0-1,Life expectancy of more than 12 weeks;
* No treated with molecular targeted drugs;
* Main organs function is normal;
* Patients should participate in the study voluntarily and sign informed consent;

Exclusion Criteria:

* Allergic to anlotinib and/or its excipients;
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure >140 mmHg，diastolic pressure>90 mmHg);
  2. Patients with Grade 2 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥450ms for male， QT≥470ms for female) and patients with Grade 3 or higher congestive heart failure (NYHA Classification) or LVEF<50%;
* Patients with a clear Gastrointestinal bleeding tendency include the following situations: Local active ulcer lesions, and fecal occult blood (+ +) ; The patient had a history of black and hematemesis within 2 months;
* Patients with a bleeding tendency and INR>1.5,APTT>1.5 ULN ;
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.);
* Patients with active brain metastasis, cancerous meningitis, spinal cord compression patients or found in Screening stage;
* Patients treated with VEGFR inhibitor;
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders;
* Patients participated in other anticancer drug clinical trials within 4 weeks;
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | up to 24 months
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm.
Disease Control Rate (DCR) | up to 24 months
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR
  + PR + SD)

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months
  The time from treatment initiation until death from any reason
Objective Response Rate (ORR) | up to 24 months
  The proportion of patients with a confirmed complete response or partial response on two consecutive occasions≥4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Quality of life score | up to 24 months
  Each 42 days up to intolerance the toxicity or PD
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 24 months
  Until initiation of new anticancer treatment
NGS(Next Generation Sequencing) detecting | up to 12 months
  The sample for NGS detecting can be gotten form storage tumor tissue specimens. It must be better collecting the new tumor tissue specimens after tumor progress

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China